CLINICAL TRIAL: NCT02651129
Title: Assessment of Noise in BC Women's Hospital Operating Rooms
Brief Title: BC Women's Hospital Noise Pilot
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Collaborators: University of British Columbia School of Population and Public Health (Unknown)
Responsible Party: Sponsor
Other Study IDs: H15-03259
Record Dates: First submitted 2015-12-18; First posted 2016-01-08 (Estimated); Last update posted 2016-11-17 (Estimated); Status verified 2016-11

CONDITIONS: Noise Levels
Keywords: noise; obstetric; operating rooms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Noise measurement — We will be measuring noise levels in the operating room

SUMMARY:
The effect of noise is often underestimated but it is one of the most common occupational health hazards. Its health effects include; noise-induced hearing loss, sleep disturbance, interference with speech comprehension, complaints, stress, annoyance, and safety concerns with regard to workers being able to complete their tasks in a safe manner.

This pilot aims to measure and analyze noise levels in obstetric ORs at BC Women's Hospital during elective and emergency cesarean deliveries.

DETAILED DESCRIPTION:
This is a pilot study that aims to measure and analyze noise levels in obstetric ORs at BC Women's Hospital during elective and emergency cesarean deliveries.

The investigators want to quantify the amount of noise in BCW ORs in order to create a research question for a larger study.

ELIGIBILITY:
Inclusion Criteria:

* BCW staff members
* Presence in OR during Cesarean section
* Willing to have a personal dosimeter pinned to hospital scrubs lapel

Exclusion Criteria:

- unable to read and understand English for the purpose of informed consent and perioperative communication

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Operating room staff
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2016-01; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
noise levels in decibels (dBs) | 1.5 hours
  during cesarean section

CONTACTS AND LOCATIONS:
Overall Officials: Vit Gubka, MD FRCPC, Principal Investigator — University of British Columbia
Locations (1):
- BC Women's Hospital, Vancouver, British Columbia, Canada